CLINICAL TRIAL: NCT02381041
Title: Comparative Evaluation of Cocaine and Adrenaline as Topical Vasonconstrictor Agents in Cosmetic Rhinoplasty
Status: Completed | Type: Observational
Sponsor: Clínica Fernández (Other)
Responsible Party: Sponsor
Other Study IDs: CF-00115-vs
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Rhinoplasty; MeSh E02.218.755
Keywords: Rhinoplasty; Topical Vasonconstrictor; Cocaine; Adrenaline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to compare two vasoconstrictive agents topically applied in cosmetic rhinoplasty: cocaine HCl 5% and adrenaline 1:1000. Blood loss during surgery as well as systemic effect of the studied agents are evaluated.

DETAILED DESCRIPTION:
A prospective non-randomized study is conducted. Female patients undergoing cosmetic rhinoplasty are included in the study.

All procedures are performed by two surgeons, both with more than ten years of experience in cosmetic rhinoplasties. One surgeon uses cocaine as the vasoconstrictor agent of choice in his daily practice, whilst adrenaline is the preferred option for the other. Both practitioners participate in all surgeries, one of them as main surgeon and the other as assistant alternatively until the study is concluded.

Vasoconstrictor effect of cocaine and adrenaline will be assessed by quantitative and qualitative evaluation. Blood loss is quantified by measuring blood aspiration during surgery and gauze weighing. Aspiration is collected in a graduated bottle; at the end of surgery fourty cc of saline is flushed through the suction system. Difference of ribbon gauze weights before and after the procedure is also measured. Adding the previous measurements gives an estimate in blood loss. Qualitative analysis of vasoconstrictive effect is based on evaluation of surgical field by each surgeon using a linear scale of 1 to 5 (1 poor, 5 excellent).

Systemic effect of vasoconstrictor drugs is assessed by heart rate (HR) and systolic/diastolic blood pressure (SBP/DBP) variations during the procedure. Patients are monitored with continuous electrocardiogram tracing and automated blood pressure. Once cocaine or adrenaline packs are placed, measurements are taken every two and a half minutes during the first ten minutes and thereafter every five minutes until the end of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Provide written consent authorization.
* Preoperatively assessed as ASA l or ll.

Exclusion Criteria:

* Known allergy to any ester based anesthetics.
* Pregnant or nursing mother.
* Any alteration of nasal mucouse that might interfere either with absorption of topical vasoconstrictor agents or with the normal wound healing process.
* Patient has used acetylsalicylic acid or NSAID 5 days prior to surgery including: ibuprofen, diclofenac, naproxen, diclofenac, indometacin, tolmetin.
* Has a known personal or family history of pheocromocytoma or adrenal tumor.
* The patient uses or has a prescribed need for stimulant drugs (amphetamines, ephedrine, norephedrine or pseudoephedrine).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Healthy females elegible for cosmetic rhinoplasty.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Bleeding in rhinoplasty procedures. | Primary outcome measures will be assessed during the surgical procedure, from the moment the vasoconstrictive agents are applied. This time period is an average of one hour.

SECONDARY OUTCOMES:
Blood pressure and heart rate variations during rhinoplasty. | Secondary outcome measures will be assessed during the surgical procedure, from the moment the vasoconstrictive agents are applied. This time period is an average of one hour.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Fernández, Oviedo, Principality of Asturias, Spain